CLINICAL TRIAL: NCT05767268
Title: Assessment of the Psychophysical State During Rehabilitation Treatment With Lokomat
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: GIP919
Record Dates: First submitted 2022-10-27; First posted 2023-03-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Acquired Brain Injury; Hereditary Spastic Paraplegia
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries; Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- treated with Lokomat: Patients perform a rehabilitation treatment of 15 or 20 sessions with lokomat + 15 or 20 sessions of physiotherapy in 3 or 4 weeks as defined by the clinician. During two or three sessions they wear a wearable device Empatica E4 that measure their electrocardiographic (ECG) activity and electrodermal activity (EDA). They also have a baseline acquisition of these signals in their room at hospital.
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — gait rehabilitation

SUMMARY:
The use of robotic technologies in rehabilitation is an increasingly widespread practice in the health sector: the Lokomat is a medical device intended for walking rehabilitation, consisting of an exoskeleton, a treadmill and a harness that supports the body weight and acts as a safety tool This technology is useful in the rehabilitation of pathologies such as prenatal stroke, brain injury, paraplegia, multiple sclerosis and other motor, orthopedic and neurological problems. During these treatments, the psychological / emotional component of the patient is not properly considered and the success of the treatment remains focused on the motor-rehabilitation level.

The management of subjective-experiential aspects remains in the hand of clinical figures (primarily physiotherapists) who have no tools for objective assessment other than their sensitivity. However, considering the experience is fundamental for the success of the therapy: this happens especially in the pediatric field, where clinical results improve significantly when children start therapy with a relaxed and positive mental state.

The aim of this project is to investigate the rehabilitation experience of patients who perform gait rehabilitation by menas of the Lokomat system, considering the relationship between physiological parameters and moods. Therefore, the main goal is to monitor the patient's psychophysical condition before, during and after the rehabilitation activity, during the different sessions. This will allow describing, with qualitative and quantitative data, the user experience of the patient who undergoes a therapeutic treatment with the Lokomat.

ELIGIBILITY:
Inclusion Criteria:

- patients that need gait rehabilitation treatment according to their clinician

Exclusion Criteria:

* subjects unable to understand and execute simple instructions;
* subjects with skin problems in the wrist area intended for the application of the Empatica bracelet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients that need gait rehabilitation treatment according to their clinician
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) session 2 | three days
  HRV is measured during the second session of Lokomat rehabilitation by means of the photoplethysmogram sensor (PPG) of Empatica E4 bracelet.
Electrodermal activity (EDA) session 2 | three days
  EDA is meadured during the second session of Lokomat rehabilitation by means of the electrodermal activity sensor of Empatica E4 bracelet.
Heart Rate Variability (HRV) session 8 | two weeks
  HRV is measured during the eighth session of Lokomat rehabilitation by means of the photoplethysmogram sensor (PPG) of Empatica E4 bracelet.
Electrodermal activity (EDA) session 8 | two weeks
  EDA is meadured during the 8th session of Lokomat rehabilitation by means of the electrodermal activity sensor of Empatica E4 bracelet.
Heart Rate Variability (HRV) session 14 | three weeks
  HRV is measured during the 14th session of Lokomat rehabilitation by means of the photoplethysmogram sensor (PPG) of Empatica E4 bracelet.
Electrodermal activity (EDA) session 14 | three weeks
  EDA is meadured during the 14th session of Lokomat rehabilitation by means of the electrodermal activity sensor of Empatica E4 bracelet.

SECONDARY OUTCOMES:
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 2 | three days
  VAS questionnaire is proposed to the subjects before the second session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.
Ad Hoc questionnaire for therapist evaluation of the patient emotional state session 2 | three days
  During the second session of Lokomat rehabilitation, the physiotherapist was asked to fill in an ad hoc questionnaire to collect a reliable evaluation of different levels of anxiety, activity, persistence of the patient. In particular, items of the proposed therapists' evaluation are reported below:
  The patient is passive/ proactive The patient is fearful/in control of the situation The patient is anxious/relaxed The patient is impulsive /thoughtful The patient is distracted /focused The patient is hyperactive/quiet The patient underestimates/overestimates his/her abilities The patient is not/ is persistent The patient is concerned/does not care about failure The patient is unable/able to derive satisfaction from success The patient manages emotions in a negative/positive manner The patient does not/does actively seek information to learn and update The therapist gives an evaluation to each item with a numerical score ranging from -3 to 3.
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 2 | three days
  VAS questionnaire is proposed to the subjects after the 8th session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 8 | two weeks
  VAS questionnaire is proposed to the subjects before the 8th session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.
Ad Hoc questionnaire for therapist evaluation of the patient emotional state session 8 | two weeks
  During the 8th session of Lokomat rehabilitation, the physiotherapist was asked to fill in an ad hoc questionnaire to collect a reliable evaluation of different levels of anxiety, activity, persistence of the patient. In particular, items of the proposed therapists' evaluation are reported below:
  The patient is passive/ proactive The patient is fearful/in control of the situation The patient is anxious/relaxed The patient is impulsive /thoughtful The patient is distracted /focused The patient is hyperactive/quiet The patient underestimates/overestimates his/her abilities The patient is not/ is persistent The patient is concerned/does not care about failure The patient is unable/able to derive satisfaction from success The patient manages emotions in a negative/positive manner The patient does not/does actively seek information to learn and update The therapist gives an evaluation to each item with a numerical score ranging from -3 to 3.
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 8 | two weeks
  VAS questionnaire is proposed to the subjects after the second session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 14 | three weeks
  VAS questionnaire is proposed to the subjects before the 14th session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.
Ad Hoc questionnaire for therapist evaluation of the patient emotional state session 14 | three weeks
  During the 14th session of Lokomat rehabilitation, the physiotherapist was asked to fill in an ad hoc questionnaire to collect a reliable evaluation of different levels of anxiety, activity, persistence of the patient. In particular, items of the proposed therapists' evaluation are reported below:
  The patient is passive/ proactive The patient is fearful/in control of the situation The patient is anxious/relaxed The patient is impulsive /thoughtful The patient is distracted /focused The patient is hyperactive/quiet The patient underestimates/overestimates his/her abilities The patient is not/ is persistent The patient is concerned/does not care about failure The patient is unable/able to derive satisfaction from success The patient manages emotions in a negative/positive manner The patient does not/does actively seek information to learn and update The therapist gives an evaluation to each item with a numerical score ranging from -3 to 3.
Ad Hoc questionnaire for patient self evaluation of his/her emotional state session 14 | three weeks
  VAS questionnaire is proposed to the subjects after the 14th session of Lokomat rehabilitation in order to collect patients' self-evaluation about their emotional state before and after the treatment.
  The following questions were proposed:
  Q1. "Are you worried?" Q2. "Are you happy" Q3. "Are you sad?" Q4. "Are you angry?" Q5. "Are you scared?" Q6. "Are you bored?" Possible answers were: not at all, a little, very much.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea, Bosisio Parini, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiappini M, Malerba G, Dei C, Bellazzecca S, Falivene A, Costantini S, Morganti R, Diella E, Storm F, Ambrosini E, Cavallo A, Biffi E. Understanding patient experience during Lokomat rehabilitation in children and adolescents: a clinical observational study combining self-evaluation and physiological metrics. BMJ Open. 2026 Feb 10;16(2):e102583. doi: 10.1136/bmjopen-2025-102583. PMID 41667181